CLINICAL TRIAL: NCT05344105
Title: Comparison of Postoperative Analgesic Efficacy of Transversalis Fascia Plan Block and Erector Spina Plan Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Hale Kefeli Celik, Principal Investigator, Anesthesiologist, Samsun Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SIMAY55
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Regional Anesthesia
Keywords: regional analgesia; transversalis fascia plane block; erector spina plane block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient will not know which study group he is in. The anesthetist, who will perform the regional block, will give the block to be applied in a sealed envelope by an assistant staff outside the study, and at the same time, the patient will not know which block has been made. The anesthesiologist who made the block will not participate in the pain follow-up of the patients. Postoperative pain assessment and data collection will be performed by another investigator blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversalis fascia plan block (Group T) (Active Comparator): After local cleaning of the skin area, the transducer will be placed on the iliac crest in the transverse plane with a low-frequency convex probe, and the skin, subcutaneous tissue, external oblique muscle will be placed with a 20 G, 100 mm needle. After visualization of the internal oblique muscle and transversus abdominis muscles and finally the deep fascia of the transversus abdominis, local anesthetic will be given unilaterally between the last part of the transversus abdominis muscle and the transversalis fascia with the out-off plan technique.
  Interventions: Device: Low frequency convex probe (ESAOTE Fixed Color Doppler Ultrasonography Device, Italy)
- Erector spina plan block (Group E) (Active Comparator): After local cleaning of the skin area, a convex probe is determined to be placed longitudinally 3 cm lateral to the spinous process of the T11 vertebra, after determining the erector spina muscle, with a 20 G, 100 mm needle inplane method in the craniocaudal direction will be advanced and a local anesthetic will be administered between the erector spinae muscle and the transverse process.
  Interventions: Device: Low frequency convex probe (ESAOTE Fixed Color Doppler Ultrasonography Device, Italy)

INTERVENTIONS:
Device: Low frequency convex probe (ESAOTE Fixed Color Doppler Ultrasonography Device, Italy) — A low frequency convex probe (ESAOTE Fixed Color Doppler Ultrasonography Device, Italy) device will be used while blocking in both groups.

SUMMARY:
The subject of the study is to compare the analgesic efficacy of transversalis fascia plan block and erector spina plane block applied with ultrasonography in patients who have undergone inguinal hernia operation. The aim of the study is to compare two different regional anesthesia methods applied in the postoperative period in terms of 24-hour opioid consumption, pain scores, additional analgesic need, and side effects and complications in the postoperative period.

DETAILED DESCRIPTION:
An identification number (ID) number will be randomly assigned to each patient, whose written consent was obtained before the surgery, when they are admitted to the postoperative recovery room. In the postoperative period, patients will be followed up with these numbers in patient follow-up. Which group the patients will be included in will be determined by the closed envelope method.

The anesthetist, who will perform the regional block, will give the block to be applied in a sealed envelope by an assistant staff outside the study, and at the same time, the patient will not know which block has been made. The anesthesiologist who made the block will not participate in the pain follow-up of the patients. Postoperative pain assessment and data collection will be performed by another investigator blinded to the study.

Spinal anesthesia will be applied to all patients and inguinal hernia operation will be appropriate. Patients taken to the recovery room will be divided into two groups. Transversalis fascia plan block (Group T) will be applied to the patients in a group after local cleansing of the skin area, accompanied by ultrasonography. The patients in the other group will be treated with an erector spina plane block (Group E) following local cleansing of the skin area, accompanied by ultrasonography.

In both block management, 0.25% bupivacaine (Buvasin Vem İlaç, Turkey) (15 ml physiological saline + 15 ml 0.5% bupivacaine) total amount of 30 ml, same volume and same concentration will be used.

After the block procedure, the patient will be observed in the recovery room for side effects. Patient-controlled analgesia (PCA) will be used as a standard in the treatment of postoperative pain in patients in both groups without any complications. Tramadol HCL, which is routinely used for postoperative pain control for PCA, will be used (3 mg/ml, total volume 100 mL).

Evaluation of postoperative pain will be done with numerical rating scale (NRS).Pain levels will be questioned in two different ways as rest and cough.

ELIGIBILITY:
Inclusion Criteria:

* Those who underwent unilateral inguinal hernia surgery under elective conditions
* 18-65 years
* ASA I-III
* Patients with written consent who agreed to participate in the study

Exclusion Criteria:

* Body mass index > 35 kg/m²,
* Coagulopathy and local infection or hematoma in the area to be blocked,
* Allergic to a local anesthetic agent or one of the drugs used in the study,
* Those with a history of chronic opioid and corticosteroid use,
* Unable to use the patient-controlled analgesia system,
* Those with psychiatric illness,
* Cases with a surgical time of less than 30 minutes and more than 120 minutes for better standardization of studies,
* Patients who do not agree to participate in the study will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Opioid use | Postoperative 24 hours
  To determine the amount of analgesic consumption in the postoperative first 24 hours with PCA in the postoperative period.

SECONDARY OUTCOMES:
Numerical Rating Scale | Postoperative 24 hours
  To determine the pain of the patients at rest and coughing at the 1st, 3rd, 6th, 12th, 18th and 24th hours postoperatively with Numerical Rating Scale (NRS).The NRS is a segmented numerical version in which the respondent selects an integer (0-10) that best reflects the intensity of their pain. 0: no pain 1-3: mild pain 4-6: moderate pain 7-10: severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Suren, Professor, Study Chair — Samsun Research and Education Hospital
Locations (1):
- Samsun Research and Education Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Researched data and statistical analyzes will be available from the journal in which the clinical study was published.

REFERENCES:
- [Result] El-Emam EM, El Motlb EAA. Ultrasound-Guided Erector Spinae versus Ilioinguinal/Iliohypogastric Block for Postoperative Analgesia in Children Undergoing Inguinal Surgeries. Anesth Essays Res. 2019 Apr-Jun;13(2):274-279. doi: 10.4103/aer.AER_81_19. PMID 31198244
- [Result] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392
- [Result] Fouad AZ, Abdel-Aal IRM, Gadelrab MRMA, Mohammed HMES. Ultrasound-guided transversalis fascia plane block versus transmuscular quadratus lumborum block for post-operative analgesia in inguinal hernia repair. Korean J Pain. 2021 Apr 1;34(2):201-209. doi: 10.3344/kjp.2021.34.2.201. PMID 33785672
- [Derived] Celik HK, Tulgar S, Buk OF, Koc K, Unal M, Genc C, Suren M. Comparison of the analgesic efficacy of the ultrasound-guided transversalis fascia plane block and erector spinae plane block in patients undergoing open inguinal hernia repair under spinal anesthesia. Korean J Anesthesiol. 2024 Apr;77(2):255-264. doi: 10.4097/kja.23404. Epub 2024 Jan 8. PMID 38185619